CLINICAL TRIAL: NCT05806164
Title: Beta-Agonist Versus OnabotulinumtoxinA Trial for Urgency Urinary Incontinence
Acronym: BEST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: University of New Mexico (Other); University of Alabama at Birmingham (Other); University of California, San Diego (Other); Howard University (Other); Brown University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Vivian Sung, MD, MPH, Professor of Obstetrics & Gynecology, The Warren Alpert Medical School of Brown University; Director of Research, Division of Urogynecology, Women & Infants Hospital of Rhode Island, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1895985
Record Dates: First submitted 2022-11-15; First posted 2023-04-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Urgency Urinary Incontinence
Keywords: UUI; Urgency Incontinence; Beta Agonist; onabotulintoxinA; Botox; Community Engagement
MeSH Terms: interventions — Adrenergic Agents; mirabegron; N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: At 3 months, the effect of treatment with beta agonist oral medication or onabotulinumtoxinA will be evaluated within a classic RCT model. The analysis will determine the effect of treatment on the co-primary outcomes: Treatment satisfaction and urinary symptom severity.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, masking of patients will not be possible; however, outcome assessors will be masked. Masked staff will not be able to see certain forms that may result in unmasking. All PROs will be administered prior to any clinical assessments to minimize bias that may occur due to clinical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta-3 receptor agonist oral medication (Active Comparator): Selective beta-3 receptor agonist oral medication approved for the treatment of urgency urinary incontinence including mirabegron or vibegron. Usual clinical care standards will be used for prescribing and dosing changes. For mirabegron, dosages are 25 mg and 50 mg as clinically indicated. For vibegron, dosage is 75 mg daily by mouth as clinically indicated.
  Interventions: Drug: Beta3-Agonists, Adrenergic [Mirabegron/Vibegron]
- Intradetrusor onabotulinumtoxinA (Active Comparator): OnabotulinumtoxinA at a dose of 100 units will be injected into the bladder per usual care pathways.
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]

INTERVENTIONS:
Drug: Beta3-Agonists, Adrenergic [Mirabegron/Vibegron] — The beta-agonist oral medication will be prescribed and dose adjusted per usual care.
  Arms: Beta-3 receptor agonist oral medication
Drug: OnabotulinumtoxinA 100 UNT [Botox] — OnabotulinumtoxinA will be prepared by dissolving 100 units into 10 ml of injectable saline. The injection will be an office based procedure, performed per usual care.
  Other Names: Botox
  Arms: Intradetrusor onabotulinumtoxinA

SUMMARY:
The goal of this clinical trial is to compare treatment outcomes between an oral medication (beta agonist) versus onabotulinumtoxinA injections in women with urgency urinary incontinence (UUI).

Participants will be randomly selected to receive one of the two treatments. The primary outcome measure will be at 3 months, and women will be followed for a total of 12 months.

Based on patient expert input, there are 2 primary outcomes: Treatment satisfaction and urinary symptom severity.

The study will also have a long-term follow-up component (prospective cohort) including 346 participants from the parent trial to describe treatment continuation, treatment efficacy, patient direct costs and other secondary outcomes up to 5 years after treatment.

DETAILED DESCRIPTION:
The purpose of this study is to directly compare 2 primary outcomes (Treatment satisfaction and urinary symptom severity) between beta agonist oral medication versus onabotulinumtoxinA intradetrusor bladder injection for the treatment of UUI.

The study will also compare secondary outcomes identified as important by patients. At the end of the study, the investigators will have patient and stakeholder-derived comparative outcomes between these 2 commonly available treatment categories. A stakeholder and community engagement (CE) plan will be developed and implemented. The investigators will also develop a model to help guide patients and providers through this decision process.

SPECIFIC AIMS Specific Aim 1: Compare the efficacy of beta agonist versus onabotulinumtoxinA on patient-important treatment outcomes at 3 months in women with UUI.

This multi-center, randomized clinical trial (RCT) includes 5 sites across the U.S. Two co-primary outcomes will be measured using validated patient-reported outcomes (PROs), selected by patients: Co-primary outcome 1: Symptom severity, measured by change in Overactive Bladder Questionnaire-Symptom Bother Scale (OAB-q-SS) score.

Co-primary outcome 2: Treatment satisfaction, measured by the Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General (FACIT-TS-G), powered based on a single item.

Specific Aim 2: Compare secondary patient-important outcomes. Direct comparisons between intervention effects on secondary outcomes chosen by patients and stakeholders, including adverse events, UUI quality of life, global improvement, and sexual function.

Specific Aim 3: Use predictive modeling to help stakeholders better determine expected outcomes after treatment with beta agonist versus onabotulinumtoxinA.

Comparators: Beta agonist oral medication (mirabegron or vibegron) versus intradetrusor onabotulinumtoxinA.

Both beta-agonists and onabotulinumtoxinA are US Food and Drug Administration (FDA) approved for the treatment of UUI, and widely available options with established efficacy.

432 women will be randomly assigned to each treatment option: 216 to beta agonist oral medication and 216 to intradetrusor onabotulintoxinA. Women will be undergo outcomes assessments at 3, 6, 9, and 12 months. The primary outcome measure will be at 3 months.

For the long-term follow up study, a prospective cohort of 346 study participants of the parent trial who agree will be followed with additional outcome assessments for 3-5 years. Outcomes for the long-term follow up study will include: continuation/discontinuation of treatment, treatment satisfaction and symptom control, treatment crossover, additional treatments, patient-important complications, costs, and understanding barriers to continued long-term UUI care and possible solutions. Qualitative methods will be expanded to further explore barriers to continuing long-term UUI care.

ELIGIBILITY:
Inclusion criteria*:

1. 18 years or older
2. report at least "quite a bit bothered" or worse by their UUI defined by response to OAB-q-SS item #8 "How bothered are you by urine loss associated with a strong desire to urinate?"
3. are not and do not plan to become pregnant
4. have persistent UUI defined as previous unsuccessful results after conservative and anticholinergic treatment, or are unable to tolerate or have contraindications to anticholinergics
5. are currently not taking anticholinergics or are willing to stop medication for 3 weeks prior to enrollment.
6. for participants reporting mixed urinary incontinence symptoms, participant must (a) have less bother from SUI than from UUI, defined as a response of "Not at all bothered" or only "a little bit bothered" by SUI on the Urogenital Distress Inventory item "Do you experience urine leakage related to physical activity? (walking, running, laughing, sneezing, coughing), and (b) SUI symptoms be stable (> 3 months), and (c)participant does not desire additional treatment for SUI in the upcoming 3 months.
7. Participants after unsuccessful neuromodulation trial can be eligible after a 4-week washout period.

Exclusion criteria:

1. clinical contraindication to beta-3 agonist or onabotulinumtoxinA
2. prior therapeutic trial of either study treatment
3. unevaluated hematuria, current or prior bladder malignancy
4. surgically altered detrusor muscle
5. prior pelvic radiation
6. post-void residual >150 mL in past 3 months
7. neurogenic bladder
8. pelvic floor surgery within the past 3 months
9. anticipating pelvic surgery within primary outcome follow up period (3 months)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in score Overactive Bladder Questionnaire-Symptom Bother Scale (OAB-q-SS) at 3 months | Baseline until 3 months
  8-item questionnaire measuring symptom bother of overactive bladder symptoms, higher scores indicate more bothersome symptoms
Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General Questionnaire (FACIT-TS-G) at 3 months | 3 months
  Single item "How do you rate this treatment overall" on a 5-point likert scale

SECONDARY OUTCOMES:
Change in Overactive Bladder Questionnaire-Symptom Bother Scale (OAB-q-SS) | Baseline until 6, 9, 12 months
  8-item questionnaire measuring symptom bother of overactive bladder symptoms
Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General Questionnaire (FACIT-TS-G) at 3 months | 6, 9, 12 months
  8-item questionnaire assessing treatment satisfaction of adults undergoing treatment for chronic conditions
Change in Overactive Bladder Questionnaire-Health Related Quality of Life (OAB-q-HRQL) | Baseline to 3, 6, 9, 12 months
  Overactive bladder disease specific questionnaire measuring quality of life, higher scores indicate better HRQL
Change in Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-IR) | Baseline to 3, 6, 9, 12 months
  Validated tool assessing female sexual function in women with pelvic floor disorders; higher scores reflect better sexual functioning
Patient global impression of improvement (PGI-I) | 3, 6, 9, 12 months
  Global measure of patient impression of improvement, likert scale

OTHER OUTCOMES:
PROMIS Cognitive Function-Short Form | Baseline to 3, 6, 9, 12 months
  Generic cognitive function measure (8 items), higher scores indicate better function
Continuation/discontinuation rate | From enrollment to end of long-term follow up 3-5 years for LTF cohort study n=346
  Continuation/discontinuation of study assigned treatment
Cost | From end of parent trial (12 months) to completion of long-term follow up study (3-5 years) for n=346
  Patient direct costs

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Sung, MD, MPH, Principal Investigator — Women and Infants Hospital of Rhode Island; Peter Jeppson, MD, Principal Investigator — University of New Mexico
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Howard University, Washington D.C., District of Columbia
  - University of New Mexico, Albuquerque, New Mexico
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The de-identified database once cleaned will be available to the team, collaborators, and broader scientific community once the primary paper is published per PCORI recommendations.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Once aims of original protocol are completed